CLINICAL TRIAL: NCT06378697
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Study to Evaluate the Efficacy and Safety of AK111 in the Treatment of Subjects With Active Ankylosing Spondylitis
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of AK111 in Subjects With Active Ankylosing Spondylitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK111-303
Record Dates: First submitted 2024-03-01; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK111 (Experimental): AK111 150 mg will be administered by subcutaneous injection at Week 0, 1 and 4 , followed by dosing every 4 weeks until Week 48.
  Interventions: Drug: AK111
- placebo (Placebo Comparator): Placebo+AK111 placebo subcutaneous injection at week 0,1, 4,8 and 12 follow AK111 4-weekly thereafter until week 48.
  Interventions: Drug: Placebo+AK111

INTERVENTIONS:
Drug: AK111 — Drug: AK111 subcutaneous injection at week 0,1, 4 and 4-weekly thereafter until week 48.
  Arms: AK111
Drug: Placebo+AK111 — Placebo+AK111 placebo subcutaneous injection at week 0,1, 4,8 and 12 follow AK111 4-weekly thereafter until week 48.
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center phase III clinical study to evaluate the efficacy and safety of AK111 in the treatment of subjects with active ankylosing spondylitis.

DETAILED DESCRIPTION:
The study consists of 3 parts. Part 1 is screening period, Part 2 is Placebo control period and part 3 is Long term treatment follow-up period. The research period is 61 weeks in total.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged ≥18 years old.
* Subjects with confirmed ankylosing spondylitis before screening.
* During screening and before randomization, BASDAI score ≥ 4, total back pain score≥ 4.
* Subjects received at least 2 kind of non-steroidal anti-inflammatory drugs (NSAIDs), prior to randomization with an inadequate response or failure to respond, or with contraindications or intolerance to the use of NSAIDs.
* Subjects who are regularly taking NSAIDs, weak opioids or oral glucocorticoids(The daily dose should be ≤10mg prednisone or equivalent dose of glucocorticoid) as part of their AS therapy are required to be on a stable dose for at least 14 days before randomization. If the drug has been discontinued, at least 2 weeks washout period is required before randomization.
* Subjects taking methotrexate (MTX) (≤25mg/week) or Sulfasalazine (≤3g/day) are allowed to continue their medication if started at least 12 weeks prior to baseline, with a stable dose for at least 4 weeks before randomization. If the drug has been discontinued, at least 4 weeks washout period is required before randomization.
* Subjects who are able to understand and voluntarily sign the ICF and complete the study procedure.

Exclusion Criteria:

* Subjects with symptom of pain that affected the evaluation of efficacy.
* Subjects with other inflammatory diseases or autoimmune diseases except Ankylosing spondylitis (AS).
* Subjects who are using strong opioid analgesics.
* Received glucocorticoid intramuscular or intravenous injection within 2 weeks prior to randomization; Received intraarticular or paraspinal glucocorticoid therapy within 4 weeks before randomization.
* Received other antirheumatic drugs (except methotrexate, sulfasalazine), proprietary Chinese medicine or traditional Chinese medicine decoction, JAK inhibitor treatment for AS within 4 weeks before randomization.
* Received Natalizumab or other B cell or T cell modulator in the 12 months prior to randomization.
* Previous exposure to secukinumab, ixekizumab or any other biologic drug directly targeting IL-17 or IL-17 receptor.
* Received multiple tumor necrosis factor α (TNF-α) inhibitors; The eluting period of biologics received before randomization is shorter than the protocol.
* Participated in a clinical study of any other drug or medical device within 1 month (≤30 days) prior to randomization, or last received the investigational drug within 5 half-lives.
* The presence of any other systemic disease or laboratory abnormalities that the investigator has judged unsuitable for clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
the response rate of ASAS20 | week 16
  Percentage of subjects who achieve Assessment of SpondyloArthritis International Society 20% improvement (ASAS20) response at Week 16.

SECONDARY OUTCOMES:
The response rate of ASAS40 | week 16
  Percentage of subjects who achieve Assessment of SpondyloArthritis International Society 40% improvement (ASAS40) response at Week 16.
The response rate of ASAS20 | baseline to week 52
  Percentage of subjects who achieve ASAS20 response throughout the clinical trial
The response rate of ASAS40 | baseline to week 52
  Percentage of subjects who achieve ASAS40 response throughout the clinical trial
The response rate of ASAS5/6 | baseline to week 52
  Percentage of subjects who achieve ≥20% improvement in five of the six domains (ASAS5/6) response throughout the clinical trial
Change from baseline on the ASDAS-CRP | baseline to week 52
  Change from baseline on the Ankylosing Spondylitis Disease Activity Score based on CRP (ASDAS-CRP) at each visit from baseline
Change from baseline on the SF-36 PCS | baseline, week 16 and week 52
  Change from baseline on the Short-Form 36 physical component score(SF-36 PCS) at each visit from baseline
Change from baseline on the ASQoL scores | baseline, week 16 and week 52
  Change from baseline on the Ankylosing Spondylitis Quality of Life (ASQoL) scores at each visit from baseline
Treatment-emergent adverse events | baseline to week 52
  Percentage of subjects with treatment-emergent adverse events (TEAEs) during the study
Serious adverse events | baseline to week 52
  Percentage of subjects with treatment-emergent serious adverse events (SAEs) during the study
Clinically significant examination results | baseline to week 52
  Recording clinically significant examination results

CONTACTS AND LOCATIONS:
Locations (54):
- China (54):
  - 1006-The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - 1038-Anhui Provincial Hospital, Hefei, Anhui
  - 1001-Peking University Third Hospital, Beijing, Beijing Municipality
  - 1002-Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - 1042-Peking University Shougang Hospital, Beijing, Beijing Municipality
  - 1049-The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - 1027-Lanzhou University Second Hospital, Lanzhou, Gansu
  - 1005-Nanfang Hospital, Guangzhou, Guangdong
  - 1025-Guangzhou First People's Hospital, Guangzhou, Guangdong
  - 1030-Jieyang People's Hospital, Jieyang, Guangdong
  - 1008-The Seventh Affiliated Hospital, Sun Yat-sen University, Shenzhen, Guangdong
  - 1026-Shenzhen People's Hospital, Shenzhen, Guangdong
  - 1056-Zhongshan Traditional Chinese Medicine Hospital, Zhongshan, Guangdong
  - 1024-Liuzhou People's Hospital, Liuchow, Guangxi
  - 1021-The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - 1022-The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - 1034-Affiliated Hospital of Hebei University, Baoding, Hebei
  - 1012-Hebei Petro China Central Hospital, Langfang, Hebei
  - 1029-Hebei General Hospital, Shijiazhuang, Hebei
  - 1033-The First Hospital of Qiqihar, Qiqihar, Heilongjiang
  - 1045-The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - 1053-Nanyang Central Hospital, Nanyang, Henan
  - 1051-Shiyan People's Hospital, Shiyan, Hubei
  - 1031-The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - 1032-Yueyang Central Hospital, Yueyang, Hunan
  - 1011-Zhuzhou Central Hospital, Zhuzhou, Hunan
  - 1017-Changzhou NO.2 People's Hospital, Changzhou, Jiangsu
  - 1037-The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - 1004-Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - 1007-Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - 1036-Jiangsu Province Hospital, Nanjing, Jiangsu
  - 1018-Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - 1035-Wuxi People's Hospital, Wuxi, Jiangsu
  - 1013-Xuzhou Central Hospital, Xuzhou, Jiangsu
  - 1014-Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - 1047-The First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - 1020-The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - 1039-The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - 1046-Pingxiang People's Hospital, Pingxiang, Jiangxi
  - 1044-Jilin Provincial People's Hospital, Changchun, Jilin
  - 1028- Jining First People's Hospital, Jining, Shandong
  - 1019-Linyi City People Hospital, Linyi, Shandong
  - 1055-Weifang People's Hospital, Weifang, Shandong
  - 1016-Zaozhuang Municipal Hospital, Zaozhuang, Shandong
  - 1054-Linfen Central Hospital, Linfen, Shanxi
  - 1009-Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - 1043-Yuncheng Central Hospital, Yuncheng, Shanxi
  - 1010-West China Hospital,Sichuan University, Chengdu, Sichuan
  - 1048-Mianyang Central Hospital, Mianyang, Sichuan
  - 1041-Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - 1023-The People's Hospital of Xinjiang Uyghur Autonomous Region, Ürümqi, Xinjiang
  - 1040- Huzhou Third People's Hospital, Huzhou, Zhejiang
  - 1015-Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - 1050-The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No